CLINICAL TRIAL: NCT05318742
Title: Panretinal Photocoagulation During Vitrectomy for Diabetic Vitreous Hemorrhage: a Randomized Clinical Trial Comparing Treatment Amount
Brief Title: Panretinal Photocoagulation During Vitrectomy for Diabetic Vitreous Hemorrhage
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Panhandle Eye Group, LLP (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Protocol 0022
Record Dates: First submitted 2022-01-01; First posted 2022-04-08 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Diabetic Vitreous Hemorrhage
MeSH Terms: interventions — Lasers

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Fewer Laser Spots (Active Comparator): Group A patients underwent endolaser PRP with a range of 200-300 shots during PPV
  Interventions: Procedure: laser
- Higher Laser Spots (Active Comparator): Group B patients underwent endolaser PRP with a range of 500-600 shots during PPV
  Interventions: Procedure: laser

INTERVENTIONS:
Procedure: laser — Endolaser photocoagulation during PPV

SUMMARY:
In this randomized clinical trial, the authors compare two cohorts receiving different endolaser spot amounts with similar laser settings in PDR subjects naïve to PRP undergoing PPV for the indication of VH.

DETAILED DESCRIPTION:
Enrolled patients will be randomized into 1 of 2 possible treatment groups: Group A patients underwent endolaser PRP with a range of 200-300 shots during PPV, whereas Group B patients underwent endolaser PRP with a range of 500-600 shots during PPV. Simple randomization will allocate subjects into treatment groups during PPV. Once all applicable maneuvers (including satisfactory hemostasis) are completed by the surgeon apart from endolaser PRP, a coin toss simulation program will randomize subjects into treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* The subject has type I or II diabetes mellitus
* The age of the subject is > 18 years old
* Snellen best-corrected visual acuity ranges from 20/40 to hand motions at one foot in the research eye
* Proliferative diabetic retinopathy with a vitreous hemorrhage is present in the research eye, and the vitreous hemorrhage is considered to be the primary cause for the subject's reduced vision
* The subject is panretinal photocoagulation-naïve
* The vitreoretinal adhesion is Grade 0 or 1 according to the classification system published by Ahn et al in the research eye

Exclusion Criteria:

* The research eye had formerly undergone anterior or posterior vitrectomy.
* An opacity of the anterior segment (cornea or lens) is thought to be responsible for two or more lines of decreased visual acuity in the research eye (cataract, corneal scar, ectasia, etc.)
* Optic nerve or retina disease unconnected to diabetes mellitus is thought to be responsible for two or more lines of decreased visual acuity in the research eye (optic neuritis, macular degeneration, glaucoma, etc.)
* Amblyopia or a non-ocular source (i.e., cerebrovascular accident) is considered to be responsible for two or more lines of decreased visual acuity in the research eye
* Neovascular glaucoma with an elevated intraocular pressure (> 30 mm Hg) is present in the research eye
* Uncontrolled systemic hypertension (systolic > 200 mmHg or diastolic > 120 mmHg) is present

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-02-15 (Actual); Primary Completion 2024-01-15 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Postoperative Vitreous Hemorrhage | 6 months
  The primary outcome measure of the trial was the incidence of postoperative VH during the 6-month trial period between treatment groups

SECONDARY OUTCOMES:
Postoperative LogMAR visual acuity | 6 months
  6 month LogMAR visual acuity between groups

CONTACTS AND LOCATIONS:
Overall Officials: Sloan Rush, MD, Study Director — panhandle eye group
Locations (1):
- La Carlota Hospital, Montemorelos, Nuevo León, Mexico

IPD SHARING:
Plan to Share IPD: No